CLINICAL TRIAL: NCT00144781
Title: A Multicenter, Multinational, Randomized, Dose-Optimization Study of the Safety and Pharmacodynamic Response of Aldurazyme® (Laronidase) in Patients With Mucopolysaccharidosis I
Brief Title: A Dose-optimization Study of Aldurazyme® (Laronidase) in Patients With Mucopolysaccharidosis I (MPS I) Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: BioMarin/Genzyme LLC (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALID-017-03
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Results first posted 2009-06-16 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Mucopolysaccharidosis I; Hurler's Syndrome; Hurler-Scheie Syndrome; Scheie Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

ARMS (4):
- 1 (Active Comparator): 0.58 mg Aldurazyme/kg of body weight (100 U/kg) administered every week (labeled dose). Final Visit is Week 27 for patients randomized to every week regimen.
  Interventions: Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase)
- 2 (Active Comparator): 1.2 mg Aldurazyme/kg of body weight (200 U/kg) administered every week. Final Visit is Week 27 for patients randomized to every week regimen.
  Interventions: Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase)
- 3 (Active Comparator): 1.2 mg Aldurazyme/kg of body weight (200 U/kg) administered every 2 weeks. Final Visit is Week 26 for patients randomized to every 2 week regimen.
  Interventions: Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase)
- 4 (Active Comparator): 1.8 mg Aldurazyme/kg of body weight (300 U/kg) administered every 2 weeks. Final Visit is Week 26 for patients randomized to every 2 week regimen.
  Interventions: Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase)

INTERVENTIONS:
Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase) — 0.58 mg/kg every week
  Arms: 1
Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase) — 1.2 mg/kg every week
  Arms: 2
Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase) — 1.2 mg/kg every other week
  Arms: 3
Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase) — 1.8 mg/kg every other week
  Arms: 4

SUMMARY:
The main purpose of this study is to evaluate differences in the pharmacodynamic response of 4 Aldurazyme® (laronidase) dose regimens in patients with Mucopolysaccharidosis I (MPS I).

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of MPS I, confirmed by measurable clinical signs and symptoms of MPS I, and a documented fibroblast or leukocyte α-L-iduronidase enzyme activity level of less than 10% of the lower limit of the normal range of the measuring laboratory.
* Weigh at least 12.5 kg.
* Have serum creatinine and blood urea nitrogen (BUN) values within age appropriate normal ranges.
* Provide signed, written informed consent prior to any protocol-related procedures being performed. Consent of a legally authorized guardian(s) is (are) required for patients under 18 years. If the patient is under 18 years old and can understand the consent, written informed consent will be required from both the patient and the authorized guardian(s).

Exclusion Criteria:

* Have previously received Aldurazyme® (laronidase).
* Have a suspected hypersensitivity to Aldurazyme® (laronidase) or known hypersensitivity to components of the infusion solution.
* Have previously undergone hematopoietic stem cell transplantation (HSCT; i.e., from bone marrow [BMT], peripheral blood, or umbilical cord blood) or other major organ transplantation.
* Have a medical condition, serious inter-current illness, or other extenuating circumstance that may interfere with study compliance including all prescribed evaluations and follow-up activities, except the 6MWT. (Note: All patients may not be capable of performing the 6MWT due to age and/or maturity level. Exemption from performing the 6MWT must be obtained in writing by the investigator from the sponsor's medical monitor prior to enrollment).
* Have an acute illness that requires surgical intervention, and/or anticipates surgery during study participation, and/or has had surgery within 30 days prior to study enrollment.
* Have received an investigational drug within 30 days prior to study enrollment.
* Is pregnant or lactating. Female patients of childbearing potential must have a negative pregnancy test [urine β-human chronic gonadotropin (hCG)] at entry (prior to the first infusion). Note: All female patients of childbearing potential and sexually mature males must be advised to use a medically accepted method of contraception throughout the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Genzyme, a Sanofi Company
Locations (5):
- Brazil (4):
  - Hospital Infantil Joana de Gusmao, Florianópolis, Santa Catarina
  - Universidade Federal de Minas Gerais, Belo Horizonte
  - Hospital de Clinical de Porto Alegre, Porto Alegre
  - Universidade Federal de Sao Paulo, São Paulo
- Division of Clinical and Metabolic Genetics, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.58 mg/kg Aldurazyme Every Week: 0.58 mg Aldurazyme/kg of body weight (100 U/kg) administered every week (labeled dose). Final Visit is Week 27 for patients randomized to every week regimen.
- 1.2 mg/kg Aldurazyme Every Week: 1.2 mg Aldurazyme/kg of body weight (200 U/kg) administered every week. Final Visit is Week 27 for patients randomized to every week regimen.
- 1.2 mg/kg Aldurazyme Every 2 Weeks: 1.2 mg Aldurazyme/kg of body weight (200 U/kg) administered every 2 weeks. Final Visit is Week 26 for patients randomized to every 2 week regimen.
- 1.8 mg/kg Aldurazyme Every 2 Weeks: 1.8 mg Aldurazyme/kg of body weight (300 U/kg) administered every 2 weeks. Final Visit is Week 26 for patients randomized to every 2 week regimen.
Period: Overall Study
Arm/Group | 0.58 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every 2 Weeks | 1.8 mg/kg Aldurazyme Every 2 Weeks
Started | 8 | 9 | 8 | 9
Completed | 8 | 7 | 8 | 9
Not Completed | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Non-compliant | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.58 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every 2 Weeks | 1.8 mg/kg Aldurazyme Every 2 Weeks | Total
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (4.86) | 8.0 (6.64) | 9.1 (4.97) | 9.3 (5.48) | 8.7 (5.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 6 | 18
  Male | 3 | 5 | 5 | 3 | 16
Study Specific Race/Ethnicity [Number; unit: participants]
  Caucasian | 4 | 6 | 5 | 6 | 21
  Black | 1 | 0 | 0 | 0 | 1
  Hispanic | 1 | 0 | 1 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0
  Other | 2 | 3 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 26 in Urinary Glycosaminoglycan (GAG) Level
Description: Urinary GAG Level - Concentration of GAG relative to creatinine in urine. A greater decrease in GAG level indicates a greater response.
Time Frame: Baseline to 26 Weeks
Population: Based on the changes in urinary GAG levels observed in the Phase 3 double-blind study, a sample size of 8 patients per group would have sufficient power to detect a 29 percentage point difference between groups in the mean change in urinary GAG levels as being statistically significant. The analysis was intention to treat.
Measure: Mean (95% Confidence Interval); unit: Percentage of Change in GAG Level
Arm/Group | 0.58 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every 2 Weeks | 1.8 mg/kg Aldurazyme Every 2 Weeks
Number analyzed (Participants) | 8 | 7 | 8 | 9
Percentage of Change in GAG Level | -57.57 (18.789) [-73.28 to -41.87] | -66.63 (14.917) [-80.42 to -52.83] | -66.15 (8.043) [-72.88 to -59.43] | -62.66 (6.506) [-67.66 to -57.66]

2. Secondary Outcome: Percent Change From Baseline to Week 26 in Liver Organ Volume
Description: A greater decrease in liver volume indicates a greater response.
Time Frame: Baseline to 26 Weeks
Population: The analysis was intention to treat.
Measure: Mean (95% Confidence Interval); unit: Percentage of Change in Liver Volume
Arm/Group | 0.58 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every 2 Weeks | 1.8 mg/kg Aldurazyme Every 2 Weeks
Number analyzed (Participants) | 7 | 7 | 8 | 8
Percentage of Change in Liver Volume | -26.27 (7.85) [-33.52 to -19.10] | -30.67 (8.13) [-38.19 to -23.15] | -30.74 (18.24) [-45.99 to -15.48] | -32.14 (10.10) [-40.58 to -23.70]

3. Secondary Outcome: Change From Baseline to Week 26 in Six Minute Walk Test (6MWT)
Description: Six Minute Walk Test: Distance walked (measured in Meters) in 6 minutes. A longer distance indicates a greater response.
Time Frame: Baseline to 26 Weeks
Population: The analysis was intention to treat.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | 0.58 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every Week | 1.2 mg/kg Aldurazyme Every 2 Weeks | 1.8 mg/kg Aldurazyme Every 2 Weeks
Number analyzed (Participants) | 6 | 6 | 7 | 7
meters | 7.00 (83.355) [-80.48 to 94.48] | -12.17 (58.043) [-73.08 to 48.75] | 25.43 (75.496) [-44.39 to 95.25] | 52.14 (72.804) [-15.19 to 119.48]

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- Aldurazyme|Every Other|Week 1.2 mg/kg***Check Title***: Aldurazyme|Every Other|Week 1.2 mg/kg***Check Description***
- Aldurazyme|Every Other|Week 1.8 mg/kg***Check Title***: Aldurazyme|Every Other|Week 1.8 mg/kg***Check Description***
- Aldurazyme|Weekly|0.58 mg/kg***Check Title***: Aldurazyme|Weekly|0.58 mg/kg***Check Description***
- Aldurazyme|Weekly|1.2 mg/kg***Check Title***: Aldurazyme|Weekly|1.2 mg/kg***Check Description***
Arm/Group | Aldurazyme|Every Other|Week 1.2 mg/kg***Check Title*** | Aldurazyme|Every Other|Week 1.8 mg/kg***Check Title*** | Aldurazyme|Weekly|0.58 mg/kg***Check Title*** | Aldurazyme|Weekly|1.2 mg/kg***Check Title***
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/9 | 1/8 | 2/8
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 8/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldurazyme|Every Other|Week 1.2 mg/kg***Check Title*** (N=8) | Aldurazyme|Every Other|Week 1.8 mg/kg***Check Title*** (N=9) | Aldurazyme|Weekly|0.58 mg/kg***Check Title*** (N=8) | Aldurazyme|Weekly|1.2 mg/kg***Check Title*** (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abasia (General disorders) | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldurazyme|Every Other|Week 1.2 mg/kg***Check Title*** (N=8) | Aldurazyme|Every Other|Week 1.8 mg/kg***Check Title*** (N=9) | Aldurazyme|Weekly|0.58 mg/kg***Check Title*** (N=8) | Aldurazyme|Weekly|1.2 mg/kg***Check Title*** (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
White blood cell disorder (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 2 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Strabismus (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 6 | 6
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 4 | 4
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Perianal erythema (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Teething (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3 | 6
Abasia (General disorders) | 0 | 0 | 1 | 0
Application site dermatitis (General disorders) | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 1
Catheter site rash (General disorders) | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1
Hernia obstructive (General disorders) | 0 | 1 | 0 | 0
Hernia pain (General disorders) | 0 | 0 | 1 | 1
Hyperthermia (General disorders) | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 2 | 0 | 2 | 3
Infusion site pruritus (General disorders) | 0 | 0 | 0 | 1
Infusion site rash (General disorders) | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 2 | 1
Pyrexia (General disorders) | 5 | 4 | 6 | 5
Vessel puncture site reaction (General disorders) | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 2 | 0
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 1 | 1 | 0
Enterobiasis (Infections and infestations) | 1 | 0 | 0 | 0
Flea infestation (Infections and infestations) | 0 | 0 | 1 | 0
Genital candidiasis (Infections and infestations) | 1 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Infection parasitic (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 3 | 2 | 1
Lice infestation (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5 | 2 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1
Otitis media acute (Infections and infestations) | 1 | 2 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 2 | 2 | 3
Sinusitis (Infections and infestations) | 4 | 2 | 2 | 3
Streptococcal impetigo (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 3
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 3 | 2 | 0 | 1
Platelet count increased (Investigations) | 1 | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Pica (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 2 | 4
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 1
Inappropriate affect (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Genital erythema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 2
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Milia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 1
Poor venous access (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study is limited by its small sample size and ability to detect small differences in urinary GAG levels between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.